CLINICAL TRIAL: NCT01167751
Title: Autologous Bone Marrow Derived Ac 133+ and Mono Nuclear Cells In-patient With Acute Myocardial Infarction During Coronary Artery Bypass Grafting (CABG): A Randomized Phase III Clinical Trial
Brief Title: Autologous Bone Marrow Derived Stem Cells for Acute Myocardial Infarction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Royan-Heart-001
Record Dates: First submitted 2010-07-19; First posted 2010-07-22 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2010-07

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Bone marrow stem cells; AC133
MeSH Terms: conditions — Myocardial Infarction | interventions — AC133 Antigen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MNC implantation (Experimental): Implantation of BM derived MNC
  Interventions: Biological: MNC
- AC 133 implantation (Experimental): Implantation of BM derived AC 133
  Interventions: Biological: AC 133
- Control (Placebo Comparator): Injection of cell carrier
  Interventions: Biological: Control

INTERVENTIONS:
Biological: MNC — Implantation of BM derived MNC
  Other Names: MNC injection
  Arms: MNC implantation
Biological: AC 133 — Implantation of BM derived AC133
  Other Names: AC133 injection
  Arms: AC 133 implantation
Biological: Control — Injection of cell carrier
  Other Names: Placebo
  Arms: Control

SUMMARY:
One of the important reasons for human dying is Ischemic heart disease (IHD). The most reason is coronary artery disease. Beside morbidity, IHD induce myocardial infarction and necrosis which due to congestive heart failure.

One therapeutic method is cellular cardiomyoplasty, which is to produce and substitute the cardiac cells with stem cell transplantation. Cell therapy is a potential therapeutic method to prevent ventricular remodeling after acute myocardial infarction. Human and animal studies have shown that stem cell trans plantation to myocardial infarcted zone can improve heart contractile function.

The aim of this study is to comparison the effects of BM-derived AC133 and MNC implantation in patients with myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* CABG candidate
* At least 4 akinetic segments
* First anterior heart attack within in 10 days to 3 month.
* St elevation MI defined by: Post Acute MI LVEF less than 45% as assessed by echocardiography.
* The target lesion had to be located in the left anterior descending (LAD) section.

Exclusion Criteria:

* History of prior anterior myocardial infarction:
* History of prior CABG
* Poor echocardiography window.
* Active infection or history of recurrent infection or positive test for syphilis (RPR), hepatitis B and C (HBSAg/ Anti HBc Anti - Hcv) HIV and HTLV-l
* Documental terminal illness or malignancy.
* Previous bone marrow transplant
* Autoimmune disease (e. g Lupus, Multiple sclerosis)
* Any contraindication for bone - marrow aspiration.
* Positive pregnancy test (in women with child bearing potential)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction at rest, measured by gated SPECT | 6 months

SECONDARY OUTCOMES:
Regional contractility in the AOI / Change in LV dimensions (left ventricular end systolic diameter [LVESD], left ventricular end diastolic diameter [LVEDD]) as assessed by echocardiography | 6 months
changes in LVM index, LVEDV, LVESV | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Royan Institute; Hossein Baharvand, PhD, Principal Investigator — Royan Institute; Mohammadhassan Nasseri, MD, Principal Investigator — Baghiatollah; Nasser Aghdami, MD, PhD, Study Director — Royan Institute
Locations (1):
- Royan Institute, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Ahmadi H, Baharvand H, Ashtiani SK, Soleimani M, Sadeghian H, Ardekani JM, Mehrjerdi NZ, Kouhkan A, Namiri M, Madani-Civi M, Fattahi F, Shahverdi A, Dizaji AV. Safety analysis and improved cardiac function following local autologous transplantation of CD133(+) enriched bone marrow cells after myocardial infarction. Curr Neurovasc Res. 2007 Aug;4(3):153-60. doi: 10.2174/156720207781387141. PMID 17691968
- [Derived] Naseri MH, Madani H, Ahmadi Tafti SH, Moshkani Farahani M, Kazemi Saleh D, Hosseinnejad H, Hosseini S, Hekmat S, Hossein Ahmadi Z, Dehghani M, Saadat A, Mardpour S, Hosseini SE, Esmaeilzadeh M, Sadeghian H, Bahoush G, Bassi A, Amin A, Fazeli R, Sharafi Y, Arab L, Movahhed M, Davaran S, Ramezanzadeh N, Kouhkan A, Hezavehei A, Namiri M, Kashfi F, Akhlaghi A, Sotoodehnejadnematalahi F, Vosough Dizaji A, Gourabi H, Syedi N, Shahverdi AH, Baharvand H, Aghdami N. COMPARE CPM-RMI Trial: Intramyocardial Transplantation of Autologous Bone Marrow-Derived CD133+ Cells and MNCs during CABG in Patients with Recent MI: A Phase II/III, Multicenter, Placebo-Controlled, Randomized, Double-Blind Clinical Trial. Cell J. 2018 Jul;20(2):267-277. doi: 10.22074/cellj.2018.5197. Epub 2018 Mar 18. PMID 29633605
- See also: Related Info — http://www.royaninstitute.org